CLINICAL TRIAL: NCT00723658
Title: S0629, Observational Study of Asymptomatic Waldenstrom's Macroglobulinemia and Phase II Study of Tandem Autologous Transplant and Maintenance Treatment for Patients With Symptomatic Disease
Brief Title: S0629, Observation or Combination Chemotherapy, Bortezomib, Thalidomide, and Rituximab Followed By Two Autologous Peripheral Blood Stem Cell Transplants in Treating Patients With Waldenstrom Macroglobulinemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0629; S0629 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2008-07-26; First posted 2008-07-29 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Lymphoma
Keywords: Waldenström macroglobulinemia
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia | interventions — Rituximab; Bortezomib; Carmustine; Cisplatin; Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; Etoposide; Melphalan; Thalidomide; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation (No Intervention): Non-symptomatic patients are monitored monthly for 3 months, then every 3 months thereafter.
- Treatment (Experimental): Symptomatic pts: 2 cycles VTDPACE+R:
  dex 40 mg PO D1-4 thalid 200 mg PO D1-4 cisplatin 10 mg/m2 IV D1-4 dox 10 mg/m2 IV D1-4 cyclophos 400 mg/m2 IV D1-4 etoposide 40 mg/m2 IV D1-4 bortezomib 1.0 mg/m2 IV D1,4,8,11 ritux 375 mg/m2 IV D1,8,15 lovenox 40 mg/d SQ D1-platelets >50,000/mcl GCSF 10 mcg/kg/d IV D9-WBC <2,000/mcl apheresis >/= 20x10^6 when WBC and CD34 within normal range, up to 4 cycles
  1. st Trans: mel 200 mg/m2 IV D-1 bortezomib 1.3 mg/m2 IV D-4, -1 PBSC >/=3.0x10^6/kg CD34 cells IV D0 GCSF 5 mcg/kg/d SQ D6-WBC recovery D5NS 500 ml IV D-1 dex 40 mg/d PO D-4 to -1 ondansetron 24 mg OR granisetron 2 mg PO D-1
  2. nd Trans: BCNU 300 mg/m2 IV D-5 etoposide 200 mg/m2 IV D-5 to -2 AraC 400 mg/m2 IV D-5 to -2 mel 140 mg/m2 IV D-1 PBSC infusion >/=3.0x10^6/kg CD34 cells IV D0 GCSF 5 mcg/kg/d SQ D6-WBC recovery D5NS 150 ml/hr IV D-5 to -1 dex 40 mg/d PO D-4 to -1 ondansetron 24 mg OR granisetron 2 mg PO D-1
  Interventions: Biological: rituximab; Drug: bortezomib; Drug: carmustine; Drug: cisplatin; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: melphalan; Drug: thalidomide; Procedure: autologous-autologous tandem hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: rituximab
  Arms: Treatment
Drug: bortezomib
  Arms: Treatment
Drug: carmustine
  Arms: Treatment
Drug: cisplatin
  Arms: Treatment
Drug: cyclophosphamide
  Arms: Treatment
Drug: cytarabine
  Arms: Treatment
Drug: dexamethasone
  Arms: Treatment
Drug: doxorubicin hydrochloride
  Arms: Treatment
Drug: etoposide
  Arms: Treatment
Drug: melphalan
  Arms: Treatment
Drug: thalidomide
  Arms: Treatment
Procedure: autologous-autologous tandem hematopoietic stem cell transplantation
  Arms: Treatment
Procedure: peripheral blood stem cell transplantation
  Arms: Treatment

SUMMARY:
RATIONALE: Sometimes the cancer may not need treatment until it progresses. In this case, observation may be sufficient. Giving combination chemotherapy together with bortezomib, thalidomide, and rituximab before an autologous peripheral stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. Giving colony-stimulating factors, such as G-CSF, helps stem cells move from the bone marrow to the blood so they can be collected and stored. More chemotherapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

PURPOSE: This observational and phase II trial is studying how well giving combination chemotherapy together with bortezomib, thalidomide, and rituximab followed by two autologous peripheral blood stem cell transplants works in treating patients with Waldenstrom macroglobulinemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the progression-free and overall survival of patients with symptomatic Waldenstrom macroglobulinemia treated with bortezomib, dexamethasone, thalidomide, cisplatin, doxorubicin hydrochloride, cyclophosphamide, and etoposide (VDT-PACE) in combination with rituximab, followed by single or tandem autologous peripheral blood stem cell transplantation and maintenance therapy.
* To assess the confirmed and unconfirmed response in patients treated with this regimen.

Secondary

* To evaluate the feasibility and toxicity of this regimen in these patients.
* To correlate the time to symptom development and overall survival with standard prognostic factors and cytopenias.
* To examine the natural history of Waldenstrom macroglobulinemia.
* To identify, in a preliminary fashion, biological correlates that may relate to progression or to symptomatic disease.

OUTLINE: This is a multicenter study. Patients with asymptomatic disease at study entry proceed directly to observation. Patients with symptomatic disease at study entry proceed directly to induction therapy.

* Observation: Patients with asymptomatic disease undergo observation monthly for 3 months and then every 3 months for up to 3 years. Patients who develop symptomatic disease proceed to induction therapy within 28 days of onset of disease symptoms. Patients who continue to have asymptomatic disease after 3 years of observation are removed from the study.
* Induction therapy: Patients receive oral dexamethasone and oral thalidomide on days 1-4; cisplatin IV, doxorubicin hydrochloride IV, cyclophosphamide IV, and etoposide IV continuously on days 1-4; bortezomib IV on days 1, 4, 8, and 11; and rituximab IV on days 1, 8, and 15. Treatment repeats every 6-8 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
* Peripheral blood stem cell (PBSC) collection: Patients receive filgrastim (G-CSF) IV beginning on day 9 of course 1 of induction therapy and continuing until WBC counts are adequate for apheresis. Patients also receive G-CSF IV beginning on day 6 of course 2 of induction therapy and continuing until apheresis is complete.
* First autologous PBSC transplantation*: Beginning approximately 4-6 weeks after the completion of induction therapy, patients receive conditioning therapy comprising high-dose melphalan IV and bortezomib IV on days -4 and -1. Patients undergo autologous PBSC transplantation on day 0 NOTE: *Patients who will receive a single transplant (for medical, insurance, or other reasons) will not receive melphalan and bortezomib, but will receive conditioning with carmustine, etoposide, cytarabine, and melphalan (BEAM) and will proceed to Maintenance Therapy.
* Second autologous PBSC transplantation: Beginning approximately 56-90 days after the first transplant, patients receive conditioning therapy comprising carmustine IV over 2 hours on day -5; etoposide IV over 1 hour and cytarabine IV over 1 hour on days -5 to -2; and melphalan IV on day -1. Patients undergo autologous PBSC transplantation on day 0.
* Maintenance therapy: Beginning after platelet counts recover, patients receive bortezomib IV on days 1, 4, 8, and 11 and rituximab IV over 2 hours on day 11. Treatment repeats every 3 months for 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Waldenstrom macroglobulinemia (WM)
* Measurable disease as determined by IgM protein quantification
* Must be registered to the treatment portion of the study within 28 days of experiencing disease-related symptoms* AND must present with ≥ 1 of the following disease-related symptoms:

  * Hemoglobin ≤ 11 g/dL
  * Platelet count ≤ 100,000/mm³
  * Marked tumor mass, defined as lymphadenopathy > 2 cm, palpable hepatomegaly, splenomegaly, or significant marrow involvement (> 50%)
  * Serum albumin < 2.5 g/dL
  * Persistently elevated beta-2-microglobulin > 3.0 mg/L in the absence of renal impairment or active infections
  * Presence of B symptoms (i.e., fever, night sweats, or weight loss of > 10% from baseline)
  * Appearance of new or worsening neuropathy manifested by numbness and tingling or pain
  * Symptomatic cryoglobulinemia (i.e., Raynaud phenomenon, skin ulcers, cold urticaria, or skin necrosis)
  * Symptoms of hyperviscosity, if measured viscosity > 4 cp (i.e., new headaches, vertigo, ataxia, dizziness with or without evident causes of changes in funduscopic exam, including retinal vein engorgement, hemorrhages, or exudates)
* NOTE: *Appearance of any of the above symptoms caused by WM with no other obvious cause is a trigger for treatment initiation. Symptoms need not persist for any specified time frame.

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2 (Zubrod performance status 3 allowed provided it is based solely on morbidity due to WM)
* ANC > 1,500/mm³ (unless more marked cytopenias can be explained by marked marrow involvement or autoimmune myelosuppression)
* Serum creatinine < 3 mg/dL
* Creatinine clearance > 30 mL/min
* SGOT/SGPT < 2 times upper limit of normal
* Direct bilirubin < 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception according to the System for Thalidomide Education and Prescribing Safety (S.T.E.P.S.®) program
* Ejection fraction ≥ 50% by ECHO or MUGA scan

  * Patients with evidence of amyloidosis (i.e., periorbital perforation, proteinuria not attributable to Bence-Jones protein, unexplained arrhythmias, increased liver function tests, peripheral neuropathy, carpal tunnel syndrome, and/or macroglossia) must have an ECHO, rather than MUGA, performed to evaluate for cardiac amyloidosis (septal thickness, diastolic dysfunction, granular sparkling, or low-voltage QRS complexes)
* No myocardial infarction within the past 6 months
* No unstable angina
* No difficult-to-control congestive heart failure or cardiac arrhythmias
* No uncontrolled hypertension
* No peripheral neuropathy ≥ grade 2
* No history of multi-infarced dementia or multiple strokes
* No known hypersensitivity to boron or mannitol
* No hepatitis B or C positivity
* No HIV positivity
* No other prior malignancy within the past 5 years except for adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* At least 28 days since prior chemotherapy and/or radiotherapy and recovered
* No prior bortezomib
* No concurrent glucocorticoids unless used to control autoimmune disease associated with WM
* Concurrent participation in the Myeloma Specimen Repository study allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 3 years | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years
Response rate (complete response, very good partial response, and partial response) | 3 years
Standard prognostic factors and other potential correlates that may relate to progression, symptomatic disease, and/or survival | 3 years
Toxicity | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Gordan Srkalovic, MD, PhD, Study Chair — Sparrow Regional Cancer Center
Locations (29):
- United States (29):
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio